CLINICAL TRIAL: NCT01746199
Title: Comparative Study of Efficacy of Two Antifolates Prophylactic Strategies Against Malaria in HIV Positive Pregnant Women (MACOMBA Study)
Brief Title: Efficacy of Antifolates Against Malaria in HIV-infected Pregnant Women and the Emergence of Induced Resistance in Plasmodium Falciparum
Acronym: MACOMBA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de Bangui (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-03
Record Dates: First submitted 2012-11-30; First posted 2012-12-10 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Malaria in Pregnancy; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cotrimoxazole daily prophylaxis (Experimental): cotrimoxazole daily prophylaxis
  Interventions: Drug: cotrimoxazole daily prophylaxis
- Intermittent Preventive sulphadoxine-pyrimethamine Treatment (Active Comparator): Referent treatment given according WHO recommendations
  Interventions: Drug: sulphadoxine-pyrimethamine

INTERVENTIONS:
Drug: cotrimoxazole daily prophylaxis
  Other Names: - CTM; - Sulfamethoxazole- trimethoprime; - Bactrim®
  Arms: cotrimoxazole daily prophylaxis
Drug: sulphadoxine-pyrimethamine — Intermittent preventive sulphadoxine-pyrimethamine treatment
  Other Names: - SP; - sulfadoxine-pyrimethamine; - Fansidar®
  Arms: Intermittent Preventive sulphadoxine-pyrimethamine Treatment

SUMMARY:
Given the resistance emergence of malaria in pregnant women receiving intermittent preventive treatment with sulfadoxine-pyrimethamine (IPT-SP) and the burden of this infection among pregnant women infected by HIV it is urgent to seek a more effective alternative treatment to optimize the prevention of malaria. Cotrimoxazole (CTM), actually administered daily as a prophylactic mean to opportunistic infections for HIV infected patients, showed encouraging results in preventing malaria in pregnant women. However, these results must be confirmed by randomized trials, particularly in pregnant women.

The main objective of this clinical trial is to compare the efficacy of cotrimoxazole (CTM), administered once daily with IPT-SP (3 curative doses spaced one month) on placental parasitaemia in pregnant women infected with HIV and cluster of differentiation 4 (CD4) > 350 cells/mm3.

The main hypothesis is based on the premise that cotrimoxazole is more effective than IPT-SP for placental parasitaemia. This might be due to the higher plasma concentration of cotrimoxazole attained with daily doses. If this hypothesis is proven, cotrimoxazole could be recommended as prophylaxis for HIV-positive pregnant women, whatever their CD4+ cell count. In this study, the investigators will also test the hypothesis that the strains of Plasmodium falciparum isolated from HIV-positive pregnant women express more dhfr and dhps resistance markers.

DETAILED DESCRIPTION:
Ascertainment of HIV serological status has become a prerequisite for better prevention of malaria. Studies reported that cotrimoxazole reduces malaria episodes in adults (other than pregnant women), and in children. Furthermore, several studies showed a good clinical and parasitological response to cotrimoxazole in treated children. Therefore, preventive treatment with SP for all HIV+ patients (including pregnant women) who are receiving treatment containing cotrimoxazole is superfluous and is even contraindicated because of the increase risk of severe adverse reactions. Few studies, however, have described the efficacy of cotrimoxazole in the prevention of malaria in pregnant women, particularly in an area where the frequency of therapeutic failures with SP in cases of Plasmodium falciparum malaria is increasing.

The emergence and augmentation of the frequency of resistance of Plasmodium falciparum to SP, which has already been observed in numerous countries of sub-Saharan Africa and in the Central African Republic, challenges the short-term usefulness of this drug combination in the prevention of malaria in pregnant women. The resistance is due to accumulation of point mutations at various sites on the genes coding for dihydrofolate reductase (dhfr) and dihydropteroate synthase (dhps). The number of mutations correlates with the extent of resistance of Plasmodium falciparum to SP in vitro. In studies carried out in Bangui, the prevalence of therapeutic failure was estimated to be 23.8% after 14 days of follow-up among children with uncomplicated malaria, while the resistance of Plasmodium falciparum to pyrimethamine in vitro was reported to be 38.3%. The frequency of mutations in dhfr and dhps alleles is correlated with in vitro response of Plasmodium falciparum strains to SP.

Pregnancy and HIV infection increase the risk for emergence of mutated strains that are resistant to SP, because a wide variety of types and clones are found in parasitaemia in pregnant women (genetic diversity). Furthermore, some studies raised concern about the possible development of cross-resistance of Plasmodium falciparum to both cotrimoxazole and SP because of the similarity of their mode of action, although this hypothesis has not been proven.

The national malaria programme in the Central African Republic recommends the use of IPT-SP since 2006.

The investigators' main hypothesis is based on the premise that cotrimoxazole is more effective than SP for placental parasitaemia. This might be due to the higher plasma concentration of cotrimoxazole attained with daily doses. If this hypothesis is proven, cotrimoxazole could be recommended as prophylaxis for HIV+ pregnant women, whatever their CD4+ cell count. In this study, the investigators will also test the hypothesis that the strains of Plasmodium falciparum isolated from HIV+ positive pregnant women express more dhfr and dhps resistance markers.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* HIV positivity
* gestational age between 16 and 28 weeks
* CD4+ count > 350 cells/mm3 and no sign of WHO stage 2, 3 or 4;
* agreement to attend all the antenatal consultations for the study
* willingness to adhere to all requirements of the study (including HIV-1 voluntary counseling and testing)
* signed informed consent

Exclusion Criteria:

* psychological instability that could interfere with compliance;
* hypersensitivity to sulfamides or dermatological disease(eczema, pemphigoid exanthema) that would increase the risk for severe reactions to the drugs being tested
* severe anaemia (Hb<7 g/dl)and any other severe disease
* known hepatic cardiac or renal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
placental parasitaemia | at parturition
  microscopic observation and confirmation by Polymerase Chain Reaction (PCR)

SECONDARY OUTCOMES:
observance CTM prophylaxis | until the end of pregnancy
occurrence of specific events related to the effectiveness of CTM prophylaxis and IPT-SP | until the end of pregnancy
  considered events :
  * maternal anemia (hemoglobinemia < 10g/dl)
  * incidence of malaria episodes during pregnancy
  * abortions, stillbirth, premature (birth <37 weeks of amenorrhea) and low birth weight (< 2500g)
  * placenta malaria and umbilical malaria transmission
occurence of adverse events | until the end of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Vray, Study Director — Unité d'épidémiologie des maladies émergentes, Institut Pasteur Paris, France; Alexandre Manirakiza, MD, Principal Investigator — Unité d'Epidémiologie, Institut Pasteur de Bangui, Central African Republic; Mirdad Kazanji, Study Chair — Director of the Institut Pasteur de Bangui, Central African Republic
Locations (4):
- Central African Republic (4):
  - Maternité de l'Hôpital communautaire, Bangui
  - Maternité de l'Hôpital de l'Amitié, Bangui
  - Maternité de la Gendarmerie Nationale, Bangui
  - Maternité du centre de santé des Castors, Bangui

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Manirakiza A, Sepou A, Serdouma E, Gondje S, Bata GG, Moussa S, Boulay A, Moyen JM, Sakanga O, Le-Fouler L, Kazanji M, Vray M. Effectiveness of two antifolate prophylactic strategies against malaria in HIV-positive pregnant women in Bangui, Central African Republic: study protocol for a randomized controlled trial (MACOMBA). Trials. 2013 Aug 14;14:255. doi: 10.1186/1745-6215-14-255. PMID 23945130